CLINICAL TRIAL: NCT01405664
Title: A Randomized, Controlled Clinical Trial to Evaluate the Effect on Patient Outcomes of Weight Bearing Status After Forage of Osteochondral Defects of the Ankle
Brief Title: the Effect of Weight Bearing Status on Healing and Pain Outcomes After Surgery for Osteochondral Defects of the Ankle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBOCD
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2022-03

CONDITIONS: Osteochondritis Dissecans of Ankle and Joints of Foot
MeSH Terms: interventions — Weight-Bearing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Weight Bearing x 6 weeks (No Intervention)
- Immediate Weight-Bearing as Tolerated (Experimental)
  Interventions: Other: Weight-Bearing as Tolerated

INTERVENTIONS:
Other: Weight-Bearing as Tolerated — WBAT immediately after surgery
  Other Names: Weight-bearing status
  Arms: Immediate Weight-Bearing as Tolerated

SUMMARY:
The rationale for this research study is to evaluate the effect on clinical outcomes of weight bearing as tolerated after forage surgery for the treatment of osteochondral defects of the ankle, thus potentially eliminating the need for a period of immobilisation or non-weight bearing after surgery.

The investigators hypothesize that their will be no difference in functional outcomes between weight bearing as tolerated as compared to non-weight bearing for six weeks after forage surgery for OCD of the ankle.

DETAILED DESCRIPTION:
The hypothesis for advantage of the investigational post-operative therapy is based on:

Equivalent clinical outcomes to non-weight bearing; Similar radiographic findings on CT at follow-up visit between the two groups; reduced morbidity and disability to subjects through elimination of a period of non-weight bearing; reduction of cost to patients by eliminating need for adjuvant walking and mobility aids (crutches, taxis) and time off work.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16-60 years
* No prior ankle surgery
* Able and willing to comply with follow-up
* Capable of provide informed consent
* Medically fit for surgery
* Lesions on preoperative CT Scan < 1.5cm
* Symptomatic (ie:pain, restricted activities, inability to WB, decreased ROM)
* Single Isolated lesion
* Failure of conservative treatment (3 months of limited activities and/or weight bearing and/or immobilization)

Exclusion Criteria:

Age less than 16 years or greater than 60 years

* Inflammatory arthritis
* Diffuse osteoarthritis of affected joint
* Associated fracture
* Prior ankle surgery for current injury (including arthroscopy)
* Unable to comply with follow-up
* Unable to provide informed consent
* Bernt & Hardy class IV (amenable to ORIF)
* Multiple osteochondral defects in one ankle or touching osteochondral lesions of tibia and talus
* Prior osteochondral defects of the affected ankle

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Ankle Osteoarthritis Scale | 12 months
  Pain and disability outcomes assessed on scale of 1-100. The higher the score is more pain\disability

SECONDARY OUTCOMES:
CAT Scan | 12months
  For assessment of cartilage healing

CONTACTS AND LOCATIONS:
Overall Officials: Mark Glazebrook, MD,FRCSC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax Infirmary, Halifax, Nova Scotia, Canada